CLINICAL TRIAL: NCT03917225
Title: A Double-Blind, Placebo-controlled Study on the Effects of MIN-102 on Biochemical, Imaging, Neurophysiological, and Clinical Markers in Patients With Friedreich's Ataxia
Brief Title: A Clinical Study to Evaluate the Effect of MIN-102 on the Progression of Friedreich's Ataxia in Male and Female Patients
Acronym: FRAMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minoryx Therapeutics, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-2-03
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Friedreich Ataxia
Keywords: Leriglitazone; Friedreich's ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIN-102 (Experimental): MIN-102 (5-[[4-[2-[5-(1-Hydroxyethyl)-2-pyridinyl]ethoxy]phenyl]methyl]-2,4-thiazolidinedione hydrochloride (1:1)). Dosing is once daily at approximately the same time each morning throughout the entire treatment phase (48 weeks).
  Interventions: Drug: MIN-102
- Placebo (Placebo Comparator): Matches MIN-102 visually and by taste. Dosing is once daily at approximately the same time each morning throughout the entire treatment phase (48 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIN-102 — Once-daily dosing with a volume specified by the pharmacokinetic specialist to achieve the desired plasma exposure. MIN-102 oral suspension, strength 15 mg/ml.
  Arms: MIN-102
Drug: Placebo — Once-daily dosing with a volume specified by the pharmacokinetic specialist. Oral suspension.
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study on the effects of MIN-102 on Biochemical, Imaging, neurophysiological, and clinical markers in patients with Friedreich's Ataxia

DETAILED DESCRIPTION:
This study investigated whether treatment with MIN-102 was able to influence clinical, neurophysiological, and imaging parameters, as well as various peripheral and central nervous system biochemical markers related to mitochondrial dysfunction, in patients with Friedreich's ataxia (FRDA), over a period of 48 weeks in a double-blind, placebo-controlled design.

Patients were screened following written consent (and assent if the patient was a minor) at the Screening visit (V-1). Eligible patients attended a Baseline visit (V0) within a maximum of 28 days after V-1 and were randomized in a 2:1 ratio to receive an individualized starting dose of MIN-102 or placebo, which they took daily for 48 weeks. Patients received individualized starting doses based on gender and age, which were subsequently modified based on pharmacokinetic (PK) parameters obtained from blood samples at V1 to achieve a target MIN-102 exposure of 170 μg.hr/mL.

In addition to the Screening visit (V-1) and Baseline visit (V0), patients were evaluated at 2 interim safety visits (ISV) occurring 2 and 8 weeks after V0 (ISV1 and ISV2; permitted to be home visits performed by a Good Clinical Practice [GCP]-certified nurse), and at 4 weeks (V1), 12 weeks (V2), 24 weeks (V3), 36 weeks (V4), and 48 weeks (V5) after V0.

Results of all scheduled assessments were made available to the investigator as soon as possible. Patients received regularly scheduled phone calls at 6, 10, 16, 20, 28, 32, 40, and 44 weeks after V0 to review changes in concomitant medications and adverse events (AEs), particularly for symptoms possibly indicative of cardiac failure. A Final Follow-up Visit (FUV) took place 4 weeks after the last dose of study drug.

Evaluations consisted of imaging evaluations at V0, V3, and V5, evaluations of clinical status using the Scale for the Assessment and Rating of Ataxia (SARA), cerebellar composite functional scale (CCFS), global clinical rating scales, and patient questionnaires at V0, V3, and V5, assessment of biochemical markers in plasma at V0, V2, V3, and V5, and blood sampling for plasma levels of MIN-102 and its main metabolite (M3) at all scheduled on-site visits (except for ISV1 and ISV2). Assessments for safety and tolerability included collection of AEs, as well as electrocardiograms (ECGs), echocardiograms, and laboratory tests. Palatability was assessed at V0, V1, V2, V3, and V4. Measurements of motor evoked potentials (MEPs) and assessment of biochemical markers in cerebrospinal fluid (CSF) were optional evaluations at V0, V3, and V5. All assessments for safety, tolerability, and biochemical markers in plasma were also performed at premature discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥12 and ≤60 years, inclusive, with a genetically confirmed diagnosis of Friedreich's Ataxia.
* Be able to walk >10 meters with support (two special sticks, stroller, or accompanying person).
* Total score on the Scale for the Assessment and Rating of Ataxia (SARA) of <25.

Exclusion Criteria:

* Age of onset of disease ≥25 years.
* Higher degree of cardiomyopathy assessed by echocardiogram.
* Diabetes.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in spinal cord area cervical segment C2-C3 [mm²] | Baseline to 48 weeks
  Spinal cord area cervical segment C2-C3 area was assessed at Baseline, Week 24, and Week 48 by morphometric magnetic resonance imaging (MRI) measurements. Morphometric changes in MRI parameters are associated with measures of clinical decline. In normal disease etiology, the spinal cord exhibits an initial decrease in area, and then reaches a plateau after 7-8 years from disease onset.

SECONDARY OUTCOMES:
Change from Baseline in SARA total score at Week 48 | Baseline to 48 weeks
  The SARA is an 8-item clinical rating scale. Five of the items are scored with points between 0 and 4, gait is scored with points between 0 and 8, and stance and speech disturbance are scored with points between 0 and 6. Total maximum score is 40 indicating maximum disability. SARA was determined at Screening, Baseline, Week 24, and Week 48.
Change from Baseline in cervical spinal cord (C2-C7) in fractional anisotropy at Week 48 | Baseline to 48 weeks
  MRI diffusion tensor imaging (DTI) was used for assessments at Baseline, Week 24, and Week 48 to measure rate of disease progression.
Change from Baseline in cervical spinal cord (C2-C7) in mean, axial, and radial diffusivity (10-³ mm²/s) at Week 48 | Baseline to 48 weeks
  MRI DTI was used for assessments at Baseline, Week 24, and Week 48 to measure rate of disease progression.
Change from Baseline in spinal cord total N-acetylaspartate concentration/myo-inositol (tNAA/mIns) ratio as assessed by magnetic resonance spectroscopy (MRS) at Week 48 | Baseline to 48 weeks
  This metabolite ratio was used to measure rate of disease progression at Baseline, Week 24, and Week 48.
Change from Baseline in quantitative susceptibility mapping (QSM) for iron concentration (ppb) at Week 48 | Baseline to 48 weeks
  QSM was acquired in the cerebellum, using a gradient echo MRI sequence. It was used to quantify local tissue properties of the dentate nucleus, which reflect iron concentration. Measurements were taken at Baseline, Week 24, and Week 48.
Change from Baseline in dentate nuclei volume at Week 48 | Baseline to 48 weeks
  QSM was acquired in the cerebellum, using a gradient echo MRI sequence. It was used to quantify local tissue properties of the dentate nucleus, including estimating the volume of the dentate nucleus. Reported values were normalized by total intracranial volume (TICV) and were dimensionless. Measurements were taken at Baseline, Week 24, and Week 48.
Change from Baseline in fixel-based analysis (FBA) of the brain at Week 48: fiber density (FD) | Baseline to 48 weeks
  Diffusion metrics related to the integrity of the corticospinal tract (CST), selected brain regions, and spinal cord fibers were extracted from diffusion-weighted images. Fixel-based analyses of the CST, the superior and inferior cerebellar peduncles (SCP and ICP), the posterior limb of the internal capsule (PLIC), the superior corna radiata (SCR), and the medial lemniscus (mLEM) were summarized to determine changes to the fibers. Fiber density measured number of axons in these structures.
Change from Baseline in fixel-based analysis (FBA) of the brain at Week 48: fiber cross-section (FC) | Baseline to 48 weeks
  Diffusion metrics related to the integrity of the CST, selected brain regions, and spinal cord fibers were extracted from diffusion-weighted images. Fixel-based analyses of the CST, the SCP and ICP, the PLIC, the SCR, and the mLEM were summarized to determine changes to the fibers. Fiber cross-section measured the area of the fiber cross-section in these structures.
Change from Baseline in fixel-based analysis (FBA) of the brain at Week 48: fiber density and cross-section (FDC) | Baseline to 48 weeks
  Diffusion metrics related to the integrity of the CST, selected brain regions, and spinal cord fibers were extracted from diffusion-weighted images. Fixel-based analyses of the CST, the SCP and ICP, the PLIC, the SCR, and the mLEM were summarized to determine changes to the fibers. Fiber density and cross-section was a combination of both FD and FC in these structures.
Change from Baseline in Cerebellar Composite Functional Scale (CCFS) at Week 48 | Baseline to 48 weeks
  The CCFS is a derived score based on results of two tests which are carried out with the dominant hand: the 9-hole peg test and clicking. The 9-hole peg test measures the time it takes for the patient to place 9 pegs in holes. In the clicking test, the subject has to press 2 buttons with the index finger of their dominant hand. The buttons are mounted on a board and have to be pressed in an alternating fashion for 10 times. As an outcome, Z-scores were calculated by subtracting the expected time that was obtained from healthy controls from the time measured in the patient. CCFS was calculated as log10 (7+Z pegboard dominant hand/10 + 4*Z click dominant hand/10). The CCFS assesses the severity of cerebellar ataxia; higher scores indicate greater severity of disease.
Change from Baseline in quality of life as measured by European Quality of Life 5 Dimensions (EQ-5D-5L) at Week 48 | Baseline to 48 weeks
  The EQ-5D-5L is a patient-rated scale with 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) where patients are asked to rate themselves according to presented responses at 5 levels of severity for each dimension (level 1 indicates no problems; level 5 indicates disability). They also rate their overall health on the particular study day on a scale from 0 to 100 points, with 0 indicating the worst possible health. The outcomes are the sum of the scores of the responses on the 5 dimensions, the overall rating of health in terms of points, and an index score based on both scores. Index scores range between 0 and 1 (with higher scores indicating better quality of life).
Change from Baseline in fatigue severity scale (FSS) at Week 48 | Baseline to 48 weeks
  Patients rate their level of fatigue on the FSS by responding to 9 presented statements where a score of 1 means maximum disagreement and 7 means strongest agreement. The outcome is the sum of scores over the 9 items. Higher scores indicate greater severity of fatigue.
Change from Baseline in Activities of Daily Living subscale of Friedreich's Ataxia Rating Scale (FARS) at Week 48 | Baseline to 48 weeks
  Activities of daily living were assessed by patients using section II of the FARS. Section II contained 9 items where subjects were rated on a scale between 0 (normal function) and 4 (most severely disturbed function). The scores for the individual 9 items are added to yield the total score. A higher score indicates a greater level of disability.
Change from Baseline in Clinician Global Impression of Severity (CGI-S) at Week 48 | Baseline to 48 weeks
  The CGI-S rates the severity of illness based on a 1-7 point scale completed by the investigator, where 1 = "normal, not at all ill" and 7 = "among the most extremely-ill patients".
Assessment from Baseline in Clinician Global Impression of Improvement (CGI-I) at Week 48 | 24 weeks and 48 weeks
  The CGI-I is a tool for assessing total overall improvement as judged by the investigator that considers whether or not the improvement is entirely due to the study medication treatment. The CGI-I rates the improvement based on a 1-7 point scale, where 1 = "very much improved" and 7 = "very much worse".
Assessment from Baseline in Patient Global Impression of Improvement (PGI-I) at Week 48 | 24 weeks and 48 weeks
  The PGI-I is a tool for assessing total overall improvement as judged by the patient during study medication treatment. The PGI-I rates the improvement based on a 1-7 point scale, where 1 = "very much improved" and 7 = "very much worse".
Percentage of patients responding to palatability of study drug questions | Baseline, Week 4, Week 12, Week 24, and Week 36
  Palatability of the study drug was assessed by the patient at Baseline, Week 4, Week 12, Week 24, and Week 36 immediately after swallowing and 10 minutes after swallowing. Patients rated the taste as "Super-good", "Good", "Neutral", "Bad", and "Super-bad". Patients were also asked if they would take the study drug every day (possible responses were "Yes", "Not sure", and "No". The percentage of patients in each category was presented.
Frequency and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Adverse events were monitored from Baseline until the Final Follow-up Visit (28 days after the last dose of study drug). TEAEs were defined as AEs occurring on or after the first dose of study drug. Number of patients with AEs and SAEs graded between Grade 1 (mild) and Grade 5 (death) was presented.
Vital signs: percentage change from Baseline in body weight (kg) | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Weight measured at Baseline and all subsequent in-person visits.
Vital signs: change from Baseline in blood pressure (mmHg) | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Systolic and diastolic blood pressure measured at Baseline and all subsequent in-person visits.
Vital signs: change from Baseline in pulse rate (beats/min) | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Measured at Baseline and all subsequent in-person visits.
Vital signs: change from Baseline in body temperature (°C) | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Measured at baseline and all subsequent in-person visits.
Number of patients with abnormal, clinically significant electrocardiogram (ECG) and echocardiogram interpretations | Baseline to Final Follow-up Visit (approximately 52 weeks)
  Echocardiograms were performed at Screening, Week 4, Week 12, Week 24, Week 24, Week 48, and the Final Follow-up Visit; 12-lead ECGs were performed at Screening, Baseline (pre-dose and 3 hours post-dose), 3 hours post-dose at Week 4, Week 12, Week 24, Week 36, and at Week 48 and the Final Follow-up Visit. The number of patients with normal, abnormal not clinically significant, abnormal clinically significant, and not assessable was tabulated.
Number of patients with abnormal, clinically significant physical examination findings | Screening to Final Follow-up Visit (approximately 56 weeks)
  Body systems examined included abdomen, extremities, heart, lungs, and skin.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Durr, Principal Investigator — ICM, Groupe Hospitalier Pitié Salpêtrière, Paris, France, 75646
Locations (5):
- Hôpital Erasme-ULB, Brussels, Belgium
- ICM, Groupe Hospitalier Pitié Salpêtrière, Paris, France
- Universitätsklinikum RWTH, Aachen, Germany
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Pandolfo M, Reetz K, Darling A, Rodriguez de Rivera FJ, Henry PG, Joers J, Lenglet C, Adanyeguh I, Deelchand D, Mochel F, Pousset F, Pascual S, Van den Eede D, Martin-Ugarte I, Vila-Brau A, Mantilla A, Pascual M, Martinell M, Meya U, Durr A. Efficacy and Safety of Leriglitazone in Patients With Friedreich Ataxia: A Phase 2 Double-Blind, Randomized Controlled Trial (FRAMES). Neurol Genet. 2022 Nov 1;8(6):e200034. doi: 10.1212/NXG.0000000000200034. eCollection 2022 Dec. PMID 36524101